CLINICAL TRIAL: NCT00890318
Title: A Study in Healthy Adult Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetic Profiles of Multiple Doses of ABT-072 Used to Treat Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Cohen, MD/Study Medical Director, Abbott
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: M10-705
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-09

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — ABT-072; Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Other): Healthy volunteers, receiving daily dose of 80 mg ABT-072 or placebo, QD for 10 days; and on Study Day 11 receiving a single dose of 80 mg ABT-072 or placebo + 400 mg ketoconazole
  Interventions: Drug: ABT-072; Other: ketoconazole; Drug: Placebo
- 2 (Other): Healthy volunteers, receiving 160 mg ABT-072 or placebo, QD for 10 days.
  Interventions: Drug: ABT-072; Drug: Placebo
- 3 (Other): Healthy volunteers, receiving 320 mg ABT-072 or placebo, QD for 10 days.
  Interventions: Drug: ABT-072; Drug: Placebo

INTERVENTIONS:
Drug: ABT-072 — Powder contents from capsules mixed in an alternative vehicle, for additional information refer to Arm Description.
Other: ketoconazole — Tablet, see Arm Description for intervention information.
  Arms: 1
Drug: Placebo — Capsule or powder drug substance from the capsule mixed in an alternative vehicle, for additional information refer to Arm Description.

SUMMARY:
The purpose of this study is to determine multiple dose safety, tolerability and pharmacokinetics of ABT-072 under nonfasting conditions in healthy adult subjects, and to determine the effect of single dose administration of ketoconazole on steady state ABT-072 pharmacokinetics.

DETAILED DESCRIPTION:
Phase 1, Blinded, Randomized, Placebo-controlled Study in Healthy Adult Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetic Profiles of Multiple Doses of ABT-072

ELIGIBILITY:
Inclusion Criteria:

* Main Selection Criteria for Healthy Volunteers:

  * Subject has provided written consent.
  * Subject is in general good health.
  * If female, subject is postmenopausal for at least 2 years or surgically sterile.
  * If female, subject is not pregnant and is not breast-feeding.
  * Male or female between 18 and 55 years old, inclusive.
  * If male, subject must be surgically sterile or practicing at least 1 method of birth control.
  * Body Mass Index (BMI) is 18 to 29, inclusive.

Exclusion Criteria:

* Use of medications including over the counter and vitamines.
* Abuse of alcohol, drugs, or nicotine.
* Current diseases or disorders.
* History of cardiac disease.
* If after consideration by the investigator, for any reason, that you are unsuitable to receive ABT-072.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Analysis of pharmacokinetic results. | Study Days 1-13
Analysis of safety measures including but not limited to tabulation of adverse events, physical exam, clinical lab results (include chemistry, hematology and urine) and vital signs. | Study Days -2 through 39

SECONDARY OUTCOMES:
Analysis of single dose administration of ketoconazole on steady state ABT-072 pharmacokinetics. | Study Day 11-13

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — Abbott
Locations (1):
- Abbott Clinical Pharmaceutical Research Unit, Waukegan, Illinois, United States